CLINICAL TRIAL: NCT05520632
Title: Autism Spectrum Disorder: Brainstem Auditory Evoked Potential Findings and Behavioral Responses to Sounds
Brief Title: Autism Spectrum Disorder: BAEPs Findings and Behavioral Responses to Sounds
Status: Recruiting | Type: Observational
Sponsor: Instituto de Ciências Biomédicas Abel Salazar (Other)
Responsible Party: Sponsor
Other Study IDs: 2021.124(101.DEFI/104-CE)
Record Dates: First submitted 2022-08-22; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Evoked Potentials, Auditory, Brain Stem

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children without autism spectrum disorder: Children without autism spectrum disorder undergoing BAEP
  Interventions: Diagnostic Test: Brainstem Auditory Evoked Potentials
- Children with autism spectrum disorder: Children with autism spectrum disorder undergoing BAEP
  Interventions: Diagnostic Test: Brainstem Auditory Evoked Potentials

INTERVENTIONS:
Diagnostic Test: Brainstem Auditory Evoked Potentials — Performing Brainstem Auditory Evoked Potentials under sedation

SUMMARY:
There are many studies in the literature that study the sensory profile of children with autism spectrum disorder (ASD), which can essentially have three types of behavior: (1) Registration, (2) Seeking, (3) Sensitivity, and (4) Avoiding. However, there are few studies dedicated to the study of the sensory profile of children with autism. A child's sensory profile is closely related to the way they deal with the world and their social interaction. The existence of tools that allow the study of the behavioral response to the sounds of children with autism spectrum disorder, will allow the application of targeted therapies in the future. Therapies targeted and adjusted to each profile observed in these children will allow to attenuate these maladjusted behavioral responses, or even overcome these deficits, if there is an early and precise intervention.

DETAILED DESCRIPTION:
The objectives of this work are:

PRIMARY OBJECTIVES:

* To characterize the BAEP findings in children with ASD (case group) and compare these findings with those obtained in children matched by sex and age without suspected ASD (control group), with a special focus on the study of the following parameters:

  1. Wave I amplitude and wave V/wave I amplitude ratio (V/I ratio)
  2. Extension of the absolute latency of wave V

     With the aim of:
     * Establish and describe a possible pattern in the BAEP that characterizes children with ASD
     * To characterize the subgroup of children with ASD who present alterations in the BAEP: understand if changes in BAEPs appear in children with more severe autism, if it depends on gender, if it depends on the auditory profile.
* Characterize the Behavioral Response to Sounds of children with ASD

  1. Application and validation for Portuguese of the Auditory Behavior Questionnaire (ABQ)
  2. Application of Child Sensory Profile 2 (CSP2) With the aim of. > To characterize the audiological profile of children with ASD
* To establish, among children with ASD, a relationship between the specific findings in the BAEP and different behavioral responses to sound.

SECONDARY OBJECTIVES:

* Collect and analyze demographic data;
* Collect and analyze the personal (pre, peri and postnatal) and family history of each participant;
* Assess the degree of global development and in particular the hearing/language parameter through data collected from the Griffiths Mental Development Scale;
* Characterize ASD in terms of severity, clinician/specialty that made the diagnosis;
* Evaluate other additional parameters of the BAEP: describe the uni or bilaterality of the findings; analyze the latency of waves III and increase in interpeak intervals for waves I-III and I-V.

MATERIAL AND METHODS

1. Study design: Analytical observational case-control study
2. Participants This study will include children between 3 and 6 years of age, observed consecutively at the Otorhinolaryngology Service of the Porto University Hospital Center and the Pediatrics Service of the Northern Mother and Child Center (belonging to the Porto University Hospital Center), with a diagnosis of ASD. with indication for performing BAEP.
3. Study groups

   The sample will be divided into two groups:
   * Children with ASD (ASD Group): cases
   * Children without diagnosis or suspicion of ASD (Group without ASD): control
4. Recruitment

   All children sent/followed at the Development Consultation - Pediatrics, Pedopsychiatry or Pediatric Neurology diagnosed with ASD aged between 2 and 6 years (potential cases) and all children aged between 2 and 6 years who have BAEP appointments in the Otorhinolaryngology department (potential controls) will be sent to the principal investigator.

   Thus, a consecutive and progressive recruitment of participants will be carried out. Parents or guardians of children who meet the inclusion criteria will be asked about their availability and interest in participating in the study, explaining the purpose of the study. An Information Leaflet for Participants has been created.

   If they wanted to participate in the study after being duly informed, an Informed Consent Term is delivered and signed.

   An individual data collection sheet was also created for data collection by the researcher. Data obtained from the electronic clinical file and provided by the parents.

   The aforementioned and scheduled BAEP questionnaires will be applied.

   After performing the BAEP, a new consultation is scheduled with the parents/legal guardians, where the result of the new assessment in terms of sensory and auditory profile, as well as the results of the BAEP will be made known.

   All data collected will go into a database created for this purpose.
5. Time line

This study will be developed in 4 main stages:

1. st PHASE: Preparation phase

   * Elaboration of the Study Protocol
   * Submission of the Project to the Ethics Committee
   * Preparation of information leaflets, consents, sheet/database for data collection
   * Creation of referral routes between the Principal Investigator and the doctors dedicated to the Development Consultation - Pediatrics, who deal with children diagnosed with ASD and with the audiologists responsible for carrying out the BAEP, in order to constitute the study sample.
   * Translation and validation of the Auditory Behavior Questionnaire
2. nd PHASE: Selection of possible study patients and data collection

   * Consecutive and progressive recruitment of participants. At this stage, the parents of children who meet the inclusion and exclusion criteria will be summoned, and asked about their availability to participate in the study;
   * The respondents that make up the study will be applied;
   * Will be requested by the BAEP researcher
3. rd PHASE: Creation of a database

   * Collection of information from BAEP;
   * All information collected and recorded on the "Individual Data Collection Sheet" in phase 2 of the study will be transferred to a database.
4. th PHASE: Data analysis and interpretation of results (2 months) The researchers and statistical analysts, using the appropriate statistical tests, will proceed to the analysis of the collected data. Subsequently, an interpretation will be made of the results of the study and a comparison with existing data in the literature in order to draw up the conclusions of the study and its dissemination in Research Article format and its presentation in free communication format at scientific events. .

6. Ethical considerations

During the realization of this study, we will act according to the medical ethics requirements defined in the World Medical Association Declaration of Helsinki - Ethical Principles for Medical Research Involving Human Subjects. Thus, this project was submitted to the Ethics Committee for Health of the Porto University Hospital Center, obtaining a favorable opinion in May/2022 (2021-124 (101-DEFI/104-CE)).

ELIGIBILITY:
Inclusion Criteria:

* Case group: children diagnosed with ASD according to the DSM-V criteria (Diagnostic and Statistical Manual of Mental Disorders 5th edition) and performed by a Pediatrician, Pedopsychiatry or Pediatric Neurologist; age between 3 and 6 years at the time of the audiological assessment; children with indication for BAEP; children who reveal thresholds within the normal range in the BAEP.
* Control group: children with typical development for their age; children with indication for BAEP due to the presence of risk factors for deafness (included in the universal neonatal auditory screening program) or due to delay in language development alone requiring clarification; age between 3 and 6 years at the time of audiological examinations; children who reveal thresholds within the normal range in the BAEP.

Exclusion Criteria:

* Case group: late diagnosis of ASD (> 6 years); associated pathology, such as: neurological (epilepsy, neurodegenerative disease, severe hypoxic-ischemic encephalopathy), congenital infections (TORCH group infections) with hearing impairment, chromosomal abnormalities (Down syndrome, fragile X syndrome), neurocutaneous syndromes, endocrine disorders and metabolic disorders (phenylketonuria), cleft palate or facial malformations; active ear pathology at the time of audiological evaluation (otitis media, external auditory canal infection or malformation); increase in auditory thresholds in BAEP.
* Control group: associated pathology, such as: neurological (epilepsy, neurodegenerative disease, severe hypoxic-ischemic encephalopathy), congenital infections (TORCH group infections) with hearing loss, chromosomal abnormalities (Down syndrome, fragile X syndrome), neurocutaneous syndromes , endocrine and metabolic disorders (phenylketonuria), cleft palate or facial malformations; active ear pathology at the time of audiological evaluation (otitis media, external auditory canal infection or malformation); increase in auditory thresholds in BAEP.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All cases as children sent/followed up in the Development Consultation - Pediatrics, Pedopsychiatry or Pediatric Neurology diagnosed with ASD aged between 2 and 6 years (possible cases) and all children aged between 2 and 6 years who had scheduled PEATC in the ENT service in routine care (possible controls)
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Findings in Brainstem Auditory Evoked Potentials (BAEP) | 3 years
  Brainstem Auditory Evoked Potentials will be performed under propofol sedation. Absolute latencies (ALs) of waves I, III, and V and interpeak latencies (IPLs) I-III, III-V, and I-V were measured, as well as the amplitudes of waves I and V. These values will be compared between the group of cases (children with ASD) and controls (children without ASD). It will be evaluated whether any of these values will be persistently outside the values considered normal in children with ASD.

SECONDARY OUTCOMES:
Study of the sensory profile of children with autism spectrum disorder applying the "Child Sensory Profile 2" questionnaire | 3 years
  Application of the questionnaire "Child Sensory Profile 2" (CSP2) and determine which category stands out: (1) Registration, (2) Seeking, (3) Sensitivity, and (4) Avoiding.
  A 5-point Likert scale (1 = almost never, 2 = occasionally, 3 = Half the time, 4 = Frequently, 5 = Almost always) will be applied to each question. A standard factor score close to zero suggests a child exhibits behaviors in that factor domain that are consistent with the majority of children. A more positive standard factor score suggests the child displays more of the observed behaviors associated with that domain than other children in this sample with ASD.
  A raw score total will be obtained for each category. Scores one standard deviation or more from the mean as expressed as "More than Others" or "Less than Others". Scotes two standard deviations or more from the mean area expressed as "Much more than the Others" or "Much less than Others", respectively.
Study of the auditory profile of children with autism spectrum disorder applying the"Auditory Behavior Questionnaire" questionnaire | 3 years
  Application of the questionnaire "Auditory Behavior Questionnaire" (ABR) and determine which category stands out in terms of auditory profile: (1) Registration, (2) Seeking, (3) Sensitivity, and (4) Avoiding.
  A 5-point Likert scale (1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Very Often.
  A a score close to zero suggests a child exhibits behaviors in that factor domain that is consistent with the majority of children with ASD. If a child has a negative standard score then the behaviors are less prevalent associated with that factor domain. A more positive standard score suggests more difficulty in the specified factor and a higher prevalence of the observed behaviors for that child.

CONTACTS AND LOCATIONS:
Overall Officials: Joana Costa, Principal Investigator — Instituto de Ciências Biomédicas Abel Salazar
Locations (1):
- Instituto de Ciências Biomédicas Abel Salazar da Universidade do Porto (Abel Salazar Biomedical Sciences Institute - University of Porto), Porto, Portugal